CLINICAL TRIAL: NCT02515825
Title: Angiographic Comparison in an Observational Study of CADence (The AMBIENCE Study)
Acronym: AMBIENCE
Status: Completed | Type: Observational
Sponsor: AUM Cardiovascular, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 1217-001
Record Dates: First submitted 2015-08-03; First posted 2015-08-05 (Estimated); Results first posted 2021-03-15 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-03

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (2):
- AMBIENCE: CADence System testing followed by coronary angiogram
  Interventions: Device: CADence
- AMBIENCE plus R&R Substudy: CADence System testing for repeatibility and reproducibility (4x by 2 operators) followed by coronary angiogram
  Interventions: Device: CADence

INTERVENTIONS:
Device: CADence

SUMMARY:
This is a prospective, multi-center study to capture information on sensitivity and specificity of CADence using coronary angiogram as the gold standard, on subjects who are already scheduled for coronary angiography.

DETAILED DESCRIPTION:
CADence is an ECG and acoustic tool to assess coronary artery disease. This study's goal is to collect patient CADence information and compare it to the results of angiogram to determine performance: sensitivity and specificity. The CADence is not used to direct patient care. This is observational only.

ELIGIBILITY:
Inclusion Criteria:

* Age >40 years
* Clinical indication for coronary angiogram
* Willing and able to give informed consent

Exclusion Criteria:

* Body Mass Index (BMI) <18.5 or >40
* Prior bypass surgery or coronary stenting
* Presence of pacemaker/defibrillator
* Presence of artificial valve
* Presence of obvious cyanotic or pre-diagnosed congenital heart defect and coarctation of the aorta
* Presence of murmurs, including valve lesions, ventricular septal defects and arteriovenous fistulae
* Presence of moderate-severe valve disease
* Left Ventricular Assist Device (LVAD)
* Presence of scars on the site thorax areas
* Participation in trial within 30 days prior to collecting CADence data except participation in registry studies.
* Asthma or chronic obstructive pulmonary disease (COPD) with active wheezing
* Inability to lie in supine position
* Heart Transplant

Min Age: 41 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects already scheduled for coronary angiography who meet study inclusion and exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 101 (Actual)
Dates: Start 2016-05; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carmelo Panetta, MD, Study Chair — University of Minnesota
Locations (3):
- United States (3):
  - Heart Center Research, LLC, Huntsville, Alabama
  - MedStar Union Memorial Hospital, Baltimore, Maryland
  - St. Joseph's Hospital, Saint Paul, Minnesota

IPD SHARING:
Plan to Share IPD: No
Data will not be shared

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects >40 years of age and scheduled for clinically-indicated angiography were recruited at 3 hospitals across the US.
Groups:
- AMBIENCE Study: Participants in the initial AMBIENCE study period
- AMBIENCE Plus R & R: Participants in the AMBIENCE plus Repeatability and Reproducibility portion of the study
Period: Overall Study
Arm/Group | AMBIENCE Study | AMBIENCE Plus R & R
Started | 70 | 31
Completed | 70 | 31
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- AMBIENCE: CADence System testing followed by coronary angiogram
  CADence System: Obtain CADence data under normal conditions of use for comparison of results with those of coronary angiogram
- AMBIENCE Plus R&R Substudy: CADence System testing for repeatability and reproducibility (4x by 2 operators) followed by coronary angiogram
  CADence System: Obtain CADence data under normal conditions for comparison of results with those of coronary angiogram.
  This part of the study includes patients who are a part of the AMBIENCE study.
- Total: Total of all reporting groups
Arm/Group | AMBIENCE | AMBIENCE Plus R&R Substudy | Total
Number analyzed (Participants) | 70 | 31 | 101
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 46 | 18 | 64
  >=65 years | 24 | 13 | 37
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.14 (8.82) | 64.65 (11.14) | 63.60 (9.56)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 6 | 29
  Male | 47 | 25 | 72
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: White | 55 | 23 | 78
  Race/Ethnicity: Black or African American | 12 | 6 | 18
  Race/Ethnicity: Asian | 1 | 0 | 1
  Race/Ethnicity: Other | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Percent of Participants With Positive Agreement of CADence Device Under Normal Use Conditions as Compared to Coronary Angiograms as Accurate and Appropriate
Description: Angiographically significant stenosis was defined as 70% or greater stenosis in any major coronary artery. Percent of Participants with Positive Agreement of CADence Device Under Normal Use Conditions as Compared to Coronary Angiograms as accurate and appropriate. The study is used to determine two conditions. CADence = Positive for 70% or greater stenosis and CADence = Negative for less than 70% stenosis. The pre-specified intent of this Outcome Measure was to assess all study participants combined, irrespective of whether or not they participated in the Ambience main study or the repeatability and reproducibility sub-study.
Time Frame: 24 hours or discharge from hospital, whichever is sooner
Population: The Ambience study included a sub-study within the same population. The sub-study was to evaluate the repeatability and reproducibility of the CADence System. Repeatability refers to the ability of the same System operator to obtain the same results each time the same subject is tested with the same System at two points in time. Reproducibility refers to the ability of different operators to obtain the same results when they evaluate the same subjects with either the same or different Systems.
Measure: Count of Participants; unit: Participants
Groups:
- Patient CADence Result: CADence System testing followed by coronary angiogram
  CADence System: Obtain CADence data under normal conditions of use for comparison of results with those of coronary angiogram
- Repeatability and Reproducibility: The purpose of the study is to collect performance information regarding the use of the CADence system under normal conditions of use. Includes a 31-subject sub-study to assess the repeatability and reproducibility of the CADence system
Arm/Group | Patient CADence Result | Repeatability and Reproducibility
Number analyzed (Participants) | 101 | 31
Participants | 101 | 31

2. Secondary Outcome: Number of Participants With CADence-related Adverse Events
Time Frame: 24 hours or discharge from hospital, whichever is sooner
Population: All participants were assessed and none had adverse events
Measure: Count of Participants; unit: Participants
Groups:
- Adverse Events: There were zero reported adverse events.
Arm/Group | Adverse Events
Number analyzed (Participants) | 101
Participants
  Adverse Events | 0
  No adverse events | 101

ADVERSE EVENTS:
Time Frame: Adverse event information was only collected through study exit for each subject (1 day).
Description: All Adverse Events (AEs) and Serious Adverse Events (SAEs) associated with CADence use through discharge were recorded. Those associated with the coronary angiogram and/or subsequent interventions were not collected.
Groups:
- AMBIENCE Plus R&R Substudy: CADence System testing for repeatibility and reproducibility (4x by 2 operators) followed by coronary angiogram
  CADence System: Obtain CADence data under normal conditions of use for comparison of results with those of coronary angiogram
Arm/Group | AMBIENCE | AMBIENCE Plus R&R Substudy
All-Cause Mortality (participants affected / at risk) | 0/70 | 0/31
Serious Adverse Events (participants affected / at risk) | 0/70 | 0/31
Other Adverse Events (participants affected / at risk) | 0/70 | 0/31

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days